CLINICAL TRIAL: NCT05294614
Title: Implementation of a Psychological Online Intervention for Low to Moderate Depression in Primary Health Care: a Study Protocol
Brief Title: Implementation of a Psychological Online Intervention for Low to Moderate Depression in Primary Health Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Conselleria de Innovación, Universidades, Ciencia y Sociedad Digital. ACIF/2020/332 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: P19/00723
Record Dates: First submitted 2021-12-14; First posted 2022-03-24 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Depressive Disorder; Depressive Symptoms; Depression
Keywords: Depressive disorder; Depression; Implementation; Evidence-based intervention; Online intervention; Psychological intervention; Primary care; Health care settings
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: The general framework determined for the study design is that indicated by Hermes. A hybrid type II design, where effectiveness and implementation will be evaluated is selected. Regarding the specific design of the empirical study, a stepped wedge (SW) design will be used, which represent a variation of the clinical trials randomized by clusters. All groups receive the treatment but its initiation is done in a randomized order and the treatment is introduced to different groups in a staggered and sequential way. The duration of each phase (e.g. control and treatment), it is determined randomly for each group. The study should be considered a closed cohort, since the same participants will be evaluated over time through a series of time points defined a priori and the inclusion of new participants will not be allowed once the trial has started. sequences will be randomly assigned.
Who Masked: Participant
Masking Description: The present work should be considered as a closed cohort study, since the same participants will be evaluated over time through a series of time points defined a priori and the inclusion of new participants will not be allowed once the trial has started. The design used for this study is composed by 3 sequences (3 different starts of the treatment phase). The assignment of each of the 6 participating centers (2 per each autonomous community) to one of the 3 sequences will be randomly performed. The established sequences look like:
  A B B B B B B B B C C C C C C A A B B B B B B B B C C C C C A A A B B B B B B B B B C C C C In these sequences A represent the control phase, B the treatment phase and the C the maintenance phase.
  Participants will be masked to the information related to the sequences that they will follow. The masking will be established according to the randomization applied to each center.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A B B B B B B B B C C C C C C (Other): Considering the study design of a closed cohort study, the design of this study is composed by 3 sequences (3 different starts of the treatment phase). In this case, the following arm is established as de first arm of the study: A B B B B B B B B C C C C C C.
  In this sequence A represent the control phase, B the treatment phase and the C the maintenance phase.
  Interventions: Behavioral: "Sonreír es diveritdo" - Smiling is fun
- A A B B B B B B B B C C C C C (Other): Considering the study design of a closed cohort study, the design of this study is composed by 3 sequences (3 different starts of the treatment phase). In this case, the following arm is established as de first arm of the study: A A B B B B B B B B C C C C C.
  In this sequence A represent the control phase, B the treatment phase and the C the maintenance phase.
  Interventions: Behavioral: "Sonreír es diveritdo" - Smiling is fun
- A A A B B B B B B B B C C C C (Other): Considering the study design of a closed cohort study, the design of this study is composed by 3 sequences (3 different starts of the treatment phase). In this case, the following arm is established as de first arm of the study: A A A B B B B B B B B C C C C.
  In this sequence A represent the control phase, B the treatment phase and the C the maintenance phase.
  Interventions: Behavioral: "Sonreír es diveritdo" - Smiling is fun

INTERVENTIONS:
Behavioral: "Sonreír es diveritdo" - Smiling is fun — Smiling is Fun is an online program with the most effective psychological procedures for depression and other techniques to promote coping ability, emotional regulation and resilience along 8 modules. The modules and their aims are: 1) Motivation for change; advantages and disadvantages of changing and importance of motivation; 2) Understanding emotional problems; psychoeducational information, maintaining factors and management of medication and sleep hygiene; 3) Learning to get going; behavioural activation strategies; 4) Learning to be flexible; how interpret negative thoughts and situations in a more flexible way; 5) Learning to enjoy; importance of positive emotions and strategies to promote them; 6) Learning to live; how to identify the psychological strengths and importance of doing activities based on values and vital goals; 7) Living and learning; putting into practice the strengths identified in previous module; 8) From now on… what?; a relapse prevention module.

SUMMARY:
Implementation of a psychological online intervention for low to moderate depression in primary care settings.

DETAILED DESCRIPTION:
Depression is highly prevalent in primary care. Meta-analysis show that pharmacotherapy and psychotherapy are effective. Given the high cost of face-to-face psychotherapy, alternative procedures of psychotherapy delivery have been proposed, emphasizing the use of technologies like the Internet. Several studies demostrated the effectiveness of Internet-based psychological interventions in primary care. Once established the efficacy and cost-effectiveness, the next step is the implementation of such programs in routine clinical practise. Literature indicates that there is a gap between the validation of evidence-based interventions and their use in routine practice of around 20 years. The science of implementation has developed procedures to reduce such gap. The objective of this study is to carry out an implementation study with a hybrid design to determine the impact of the intervention (Smiling is Fun) in terms of health outcomes and feasibility of the implementation. Participants will adopt the framework proposed by Hermes et al., inspired in Proctor's recommendations. The study will be conducted in Andalucia, Aragon and Baleares. It is hypothesized that it will be feasible to implement a psychological intervention supported by ICTs in the context of primary care for the treatment of mild-moderate depression. Furthermore, specific hypothesis are established; 1) the intervention will be effective after six months of completion of treatment (efficacy measure: PHQ9), 2) the psychological intervention applied through ICTs in primary care will be cost-effective, 3) the acceptability of the intervention will be high by the agents involved: patients, professionals and administrators (results of interviews and focus groups), this acceptability will also be high with regarding the usability of the designed computer system (measured by the System Usability Scale), 4) the data about the use of the platform by patients and professionals will demonstrate that the intervention is adopted, feasible, and high fidelity (modules and tasks completed) and 5) the adequacy of the ICT-supported intervention perceived by professionals, patients andadministrators will be elevated (NoMAD questionnaire and results of interviews and focus groups).The final goal of this study is to demonstrate the feasibility of using the online intervention in order to guarantee that the investment in efficacy research lead to a better care in routine clinical practice and an improvement in public health.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18 years old.
* DSM-5 Diagnosis of Major Depression.
* Severity of mild or moderate depression (score less than 14 points on PHQ-9).
* Duration of depressive symptoms 2 months or more.
* Availability of computer with Internet connection.
* Understand Spanish spoken and written.
* Give informed consent.

Exclusion Criteria:

* Disease affecting the Central Nervous System.
* Other psychiatric diagnosis or illness severe psychiatric (substance dependence and abuse, psychosis, eating disorders, etc.) a exception of anxiety pathology or personality disorders.
* Presence of medical illness, uncontrolled severe degenerative or infectious disease.
* Presence of delusions or hallucinations in the time of study.
* Risk of suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the intervention | Pre-intervention and immediately after the intervention
  Change of depression symtpmatology through the Patient Health Questionnaire-9 (PHQ-9) after the intervention.

SECONDARY OUTCOMES:
Acceptability | Pre-intervention and immediately after the intervention
  Assesment of the usability, defined as the facility of use percibed by the users through the System Usability Scale.
Acceptability | Immediately after the intervention
  Satisfaction of the online intervention through the Client Satisfaction Questionnaire (CSQ-1).
Adaptation | Pre-intervention, immediately after the intervention and follow-up
  Assesment of the process of normalization of an intervention through the Normalization MeAsure Development Questionnaire (NoMAD).
Adoption, viability and fidelity | Pre-intervention and immediately after the intervention
  Assessed with the infromation proportioned by the online intervention. Specifically: number of access to the application, number of completed modules and number of performed tasks
Implementation costs | Pre-intervention and immediately after the intervention AND follow-up
  Assessment of the use of health and social services and other economical impacts thourgh the Client Service Receipt Inventory (CSRI).
Diagnostic Interview | Pre-intervention
  Assessment of the diagnostic criteria included in the DSM-V.

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García Palacios, Principal Investigator — University Jaume I; Javier García Campayo, Principal Investigator — Institute of Health Research of Aragon; Margalida Gili, Principal Investigator — Research Institute of Health Sciences, University of Balearic Islands, Palma de Mallorca; Fermín Mayoral Cleries, Principal Investigator — University Regional Hospital of Malaga
Locations (1):
- Rosa Lorente Català, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mira A, Soler C, Alda M, Banos R, Castilla D, Castro A, Garcia-Campayo J, Garcia-Palacios A, Gili M, Hurtado M, Mayoral F, Montero-Marin J, Botella C. Exploring the Relationship Between the Acceptability of an Internet-Based Intervention for Depression in Primary Care and Clinical Outcomes: Secondary Analysis of a Randomized Controlled Trial. Front Psychiatry. 2019 May 10;10:325. doi: 10.3389/fpsyt.2019.00325. eCollection 2019. PMID 31133899
- [Background] Romero-Sanchiz P, Nogueira-Arjona R, Garcia-Ruiz A, Luciano JV, Garcia Campayo J, Gili M, Botella C, Banos R, Castro A, Lopez-Del-Hoyo Y, Perez Ara MA, Modrego-Alarcon M, Mayoral Cleries F. Economic evaluation of a guided and unguided internet-based CBT intervention for major depression: Results from a multi-center, three-armed randomized controlled trial conducted in primary care. PLoS One. 2017 Feb 27;12(2):e0172741. doi: 10.1371/journal.pone.0172741. eCollection 2017. PMID 28241025
- [Background] Montero-Marin J, Araya R, Perez-Yus MC, Mayoral F, Gili M, Botella C, Banos R, Castro A, Romero-Sanchiz P, Lopez-Del-Hoyo Y, Nogueira-Arjona R, Vives M, Riera A, Garcia-Campayo J. An Internet-Based Intervention for Depression in Primary Care in Spain: A Randomized Controlled Trial. J Med Internet Res. 2016 Aug 26;18(8):e231. doi: 10.2196/jmir.5695. PMID 27565118
- [Background] Montero-Marin J, Prado-Abril J, Botella C, Mayoral-Cleries F, Banos R, Herrera-Mercadal P, Romero-Sanchiz P, Gili M, Castro A, Nogueira R, Garcia-Campayo J. Expectations among patients and health professionals regarding Web-based interventions for depression in primary care: a qualitative study. J Med Internet Res. 2015 Mar 10;17(3):e67. doi: 10.2196/jmir.3985. PMID 25757358
- [Background] Karyotaki E, Kemmeren L, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJH, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Is self-guided internet-based cognitive behavioural therapy (iCBT) harmful? An individual participant data meta-analysis. Psychol Med. 2018 Nov;48(15):2456-2466. doi: 10.1017/S0033291718000648. Epub 2018 Mar 15. PMID 29540243
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Mira A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos RM, Botella C. An Internet-based program for depressive symptoms using human and automated support: a randomized controlled trial. Neuropsychiatr Dis Treat. 2017 Mar 31;13:987-1006. doi: 10.2147/NDT.S130994. eCollection 2017. PMID 28408833
- [Background] Karyotaki E, Kleiboer A, Smit F, Turner DT, Pastor AM, Andersson G, Berger T, Botella C, Breton JM, Carlbring P, Christensen H, de Graaf E, Griffiths K, Donker T, Farrer L, Huibers MJ, Lenndin J, Mackinnon A, Meyer B, Moritz S, Riper H, Spek V, Vernmark K, Cuijpers P. Predictors of treatment dropout in self-guided web-based interventions for depression: an 'individual patient data' meta-analysis. Psychol Med. 2015 Oct;45(13):2717-26. doi: 10.1017/S0033291715000665. Epub 2015 Apr 17. PMID 25881626
- [Background] GBD 2015 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 315 diseases and injuries and healthy life expectancy (HALE), 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1603-1658. doi: 10.1016/S0140-6736(16)31460-X. PMID 27733283
- [Background] Pakenham-Walsh, Neil. (2004). Learning from one another to bridge the "know-do gap". BMJ. 329. 10.1136/bmj.329.7475.1189.
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Derived] Lorente-Catala R, Gili M, Lopez-Del-Hoyo Y, Mayoral-Cleries F, Perez-Aranda A, Castro A, Varela-Moreno E, Banos RM, Roca M, Monreal-Bartolome A, Garcia-Palacios A. Implementation of a psychological online intervention for low to moderate depression in primary care: study protocol. Internet Interv. 2022 Nov 1;30:100581. doi: 10.1016/j.invent.2022.100581. eCollection 2022 Dec. PMID 36573071